CLINICAL TRIAL: NCT01323127
Title: Preliminary Study of the Sagittal Alignment of the Lumbo-pelvic Complex in a Sitting Position
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2010/AD-03; 2010-A01536-33 (Other: ANSM)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Back Pain; Low Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic back pain: This group of patients has had chronic back pain for longer than 3 months.
  Interventions: Procedure: Sagital xrays
- Non chronic back pain: This group of patients is hospitalized for cardio physical therapy, and has no lumbar-pelvic complications. Patients are selected from the hospitalized population according to age, sex, and BMI in order to match chronic back pain patients.
  Interventions: Procedure: Sagital xrays

INTERVENTIONS:
Procedure: Sagital xrays — 5 xrays will be taken: (1) Upright standing position; (2) Upright, straight chair position; (3) Slouching, straight chair position; (4) Upright, ergonomic chair position; (5) Slouching, ergonomic chair position.

SUMMARY:
The main objective of this study is to investigate the influence of seat type (straight chair versus "ergonomic" chair) on the sagittal alignment of the lumbo-pelvic complex in two different postures compared to standing for each individual in both a chronic-back-pain and a non-chronic-back-pain population.

ELIGIBILITY:
General Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan

Inclusion Criteria for the Chronic Back Pain Group

* Patient has chronic lombalgia (> 3 months)
* Patient has discopathy evidenced by standard imaging of the lumbar spine

Inclusion Criteria for the Non Chronic Back Pain Group

* Patient does not have chronic lombalgia or neurological symptoms
* Patients hospitalized for cardiovascular physical therapy which does not interfere with the sagital alignment of the lombo-pelivien complex (post-infarctus care, cardiac insufficiency)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The subject has had more than two x-rays, or similar ray exposure during the previous year
* The subject has a professional activity or hobby that exposes him/her to radiation
* The subject has a lombo-pelivien malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two populations are compared: one with chronic back pain, and the other a group of hospitalized patients with no lombo-peliven complications.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12-10 (Actual); Study Completion 2011-12-10 (Actual)

PRIMARY OUTCOMES:
% variation in the pelvic incidence angle in sitting compared to standing | Upon xray; day 1

SECONDARY OUTCOMES:
% variation in the sacral slope angle in sitting compared to standing | upon xray; Day 1
% variation in the pelvic tilt angle in sitting compared to standing | upon xray; Day 1
% variation in the lumbar lardosis angle in sitting compared to standing | upon xray; Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

REFERENCES:
- [Result] Vaucher M, Isner-Horobeti ME, Demattei C, Alonso S, Herisson C, Kouyoumdjian P, van Dieen JH, Dupeyron A. Effect of a kneeling chair on lumbar curvature in patients with low back pain and healthy controls: A pilot study. Ann Phys Rehabil Med. 2015 Jun;58(3):151-6. doi: 10.1016/j.rehab.2015.01.003. Epub 2015 May 5. PMID 25956202